CLINICAL TRIAL: NCT03585634
Title: The Dads in Gear Program: An Innovative Men-centered Approach to Smoking Cessation
Acronym: DIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Joan Bottorff, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: #702831
Record Dates: First submitted 2018-05-25; First posted 2018-07-13 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Smoking Cessation
Keywords: Fathers; Masculinity; Gender role; Health Behaviour; Family health
MeSH Terms: conditions — Smoking Cessation; Masculinity | interventions — amsonic acid

STUDY DESIGN:
Intervention Model Description: Prospective, non-comparative design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dads in Gear Program (Other): An 8 week group program to support men's smoking cessation efforts.
  Interventions: Behavioral: Dads in Gear Program

INTERVENTIONS:
Behavioral: Dads in Gear Program
  Other Names: DIG program

SUMMARY:
The purpose of this feasibility study is to evaluate Dads in Gear, a tailored program to support expectant and new fathers efforts to quit smoking. The 8 week group program integrates peer support and resources to support cessation, physical activity, and knowledge and skills related to fathering.

DETAILED DESCRIPTION:
Using a prospective, non-comparative design, the DIG program is implemented and evaluated in 6 communities in this feasibility study. The program is offered by trained facilitators to fathers who currently smoke and want to quit. The RE-AIM framework is used to guide the evaluation. Open-ended questions in participant surveys, and semi-structured interviews and weekly telephone de-briefs with facilitators provide data for a process evaluation. Estimates of effectiveness include smoking behavior, fathering and physical activity measures at baseline, end of program, and 3-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Fathers of any age
* Currently smoking and want to quit smoking, or recently quit smoking (within last 2 months)
* Have at least one child under 5 years old or expecting a child (Men do not have to be residing with their children to be eligible)
* Able to attend the group program

Exclusion Criteria:

- Non smokers

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Men any age, currently smoking, want to quit smoking, recently quit smoking and have a child under 5 years old or expecting a child.
Enrollment: 36 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Change in smoking status from baseline to end of 8 week program | Baseline, and at end of 8 week program
  Self-reported smoking status using the following questions: Are you currently smoking? [Response: Yes/No]. If NO, how long have you been smoke-free? [Response: ___ # of days ___ # of weeks]
Smoking status at 3 months following end of 8 week program | 3 month follow-up
  Self-reported smoking status using the following questions: Are you currently smoking? [Response: Yes/No]. If NO, how long have you been smoke-free? [Response: ___ # of days ___ # of weeks]

SECONDARY OUTCOMES:
Smoking behaviour - quit attempts during 8 week program | End of 8 week program
  Self-reported frequency of quit attempts (smoke free for at least 24 hours) (questionnaire item)
Smoking behaviour - quit attempts between end of program and 3 month follow-up | At 3 month follow-up
  Self-reported frequency of quit attempts during previous 3 months (smoke free for at least 24 hours) (questionnaire item)
Confidence to stay smoke free at end of 8 week program | End of 8 week program
  Self-reported confidence to stay smoke free (questionnaire item)
Confidence to stay smoke free at 3 month follow-up | 3 month follow-up
  Self-reported confidence to stay smoke free (questionnaire item)
Change in Fathering Self-Efficacy from baseline to end of 8 week program | Baseline and at end of 8 week program
  Fathering Self-efficacy Scale developed by Sevigney et al. (2016) is a measure of men's perceptions of their abilities (self-efficacy) related to parenting and fatherhood. Two of the three sub-scales in this tool will be used: Positive engagement (12 items; with scores ranging from 12 - 120) and direct care (4 items, with scores ranging from 4 - 40). A 10-point Likert scale response format is used for each item. The item scores in each sub-scale will be summed to obtain sub-scale scores. Sub-scale scores are summed for total Father Self-Efficacy score (range 16-160). Higher scores indicate better self-efficacy.
Fathering Self-efficacy at 3 month follow-up | 3 month follow-up
  Fathering Self-efficacy Scale developed by Sevigney et al. (2016) is a measure of men's perceptions of their abilities (self-efficacy) related to parenting and fatherhood. Two of the three sub-scales in this tool will be used: Positive engagement (12 items; with scores ranging from 12 - 120) and direct care (4 items, with scores ranging from 4 - 40). A 10-point Likert scale response format is used for each item. The item scores in each sub-scale will be summed to obtain sub-scale scores. Sub-scale scores are summed for total Father Self-Efficacy score (range 16-160). Higher scores indicate better self-efficacy.
Change in physical activity from baseline to end of 8 week program | Baseline, and at end of 8 week program
  Godin Physical activity leisure time questionnaire
Physical activity at 3 month follow-up | 3 month follow-up
  Godin Physical activity leisure time questionnaire
Change in sedentary behavior from baseline to end of 8 week program | Baseline, and end of 8 week program
  Self-reported time spent sitting during past 7 days on a weekday (questionnaire item).
Sedentary behavior at 3 month follow-up | 3 months follow-up
  Self-reported time spent sitting during past 7 days on a weekday (questionnaire item).

OTHER OUTCOMES:
Program Fidelity | During 8 week program implementation
  Semi-structured telephone interviews with facilitators during program implementation

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bottorff, PhD, Principal Investigator — University of British Columbia; John Oliffe, PhD, Principal Investigator — University of British Columbia

REFERENCES:
- [Background] Bottorff JL, Oliffe JL, Sarbit G, Caperchione C, Clark M, Anand A, Howay K. Assessing the feasibility, acceptability and potential effectiveness of an integrated approach to smoking cessation for new and expectant fathers: The Dads in Gear study protocol. Contemp Clin Trials. 2017 Mar;54:77-83. doi: 10.1016/j.cct.2017.01.002. Epub 2017 Jan 11. PMID 28088514
- See also: Dads in Gear Website — http://dadsingear.ok.ubc.ca/